CLINICAL TRIAL: NCT04147689
Title: Evaluation of the Efficacy and Safety of Hyaluronic Acid Injection in Labia Majora for Volume Restoration
Acronym: ESOLANE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A01241-56
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Vulvar Atrophy
Keywords: hyaluronic acid; labia majora; vulvar; filler; hypotrophy; atrophy
MeSH Terms: conditions — Atrophy

STUDY DESIGN:
Intervention Model Description: One group of patient treated with DESIRIAL® PLUS (injection in labia majora)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated labia majora (Experimental): Labia majora are treated at Baseline visit (V1) and a touch-up may be performed 4 weeks after Baseline (V2) if needed
  Interventions: Device: DESIRIAL® PLUS

INTERVENTIONS:
Device: DESIRIAL® PLUS — DESIRIAL® PLUS is a cross-linked hyaluronic acid gel to restore volume by filling the labia majora, to rehydrate and to add tone and tension to the area of connective tissue.
  The baseline injection is performed at V1, with a maximum volume to be injected per labium of 2 ml. The exact volume will be determined by the physician in order to reach optimal volume correction.
  One optional touch-up injection of DESIRIAL® PLUS is allowed at V2 (4 weeks after Baseline), with a maximum volume to be injected per labium of 1 ml. No other touch-up injections are allowed until the end of the study.

SUMMARY:
DESIRIAL® PLUS is a CE-marketed hyaluronic acid (since 2011) whose registered indications are moderate hypotrophy, severe hypotrophy or atrophy of the vulvar Labia Majora by subcutaneous injections. The aim is to restore volume, rehydrate and add tone and tension to connective tissue areas by filling.

In this study, 71 female subjects above or equal to 18 years old at inclusion, who have moderate hypotrophy or severe hypotrophy or atrophy of the vulvar Labia Majora (according to investigator's judgement), who have given her informed consent and meet all the eligibility criteria, will be enrolled. Subjects will come to a total of 6 visits over a period of 12 months. An optional screening visit may be done before injection (additional visit). Proportion of patients having an improved perception of aesthetics (GAIS score after mirror self-examination) after baseline injection will be assessed. Global Aesthetic Improvement, Sexual function, subject's satisfaction, subject's symptoms, pain at injection and safety will be also assessed.

DETAILED DESCRIPTION:
ESOLANE is a prospective multicenter post-marketing study of a class III medical device. This uncontrolled open-label study investigates the efficacy and safety of DESIRIAL® PLUS in volume restoration of Labia Majora. The study duration is 12 months with an optional screening visit (V0) up to 14 days before injection, the baseline visit (injection of DESIRIAL®PLUS, V1) and 5 follow-up visits after 4, 12, 24, 36 and 52 weeks (V2 to V6). At 4 weeks (V2) an optional touch-up may be done (if needed). It is envisaged to enrol 71 female patients with the wish for volume restoration in France to obtain at least 60 evaluable patients, which will be monitored over 1 year after baseline injection of DESIRIAL® PLUS.

The primary endpoint is defined as the proportion of patients having an improved perception of aesthetics (GAIS score after mirror self-examination) at 12 weeks after baseline injection of DESIRIAL® PLUS, which may be touched-up once after 4 weeks (V2).

Global Aesthetic Improvement (evaluated by the patient and the doctor), Sexual function, subject's satisfaction, subject's symptoms & pain, will be measured at all time-point with a Global Aesthetic Improvement Scale (GAIS), Female Sexual Function Index (FSFI), patient's satisfaction questionnaire (PSQ) and a Numerical Rating Scale (NRS) respectively. Safety will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

Women with the following conditions :

* ≥ 18 years of age at inclusion
* Moderate hypotrophy, severe hypotrophy or atrophy of the vulvar Labia Majora, according to the investigator's judgement
* Expressed the wish for volume restoration of the Labia Majora
* Able to understand and sign the informed consent for study enrolment
* Subject affiliated to a health social security system

Non-inclusion Criteria

General :

* Pregnancy
* Breast feeding
* Known tendency to develop hypertrophic scars or keloid scars
* Participating at the same time in another clinical trial
* Deprived of their freedom by administrative or legal decision or under guardianship

Linked to inflammatory or immune status:

* Known hypersensitivity

  * to one of DESIRIAL® PLUS's components (hyaluronic acid, mannitol)
  * to the antiseptic solution that is planned to be used in this study
  * to amide local anesthetics or to one of the components of the anesthesia product that is planned to be used in this study
* Presence of clinical signs of inflammatory in or close to the area of interest or treatment for these affections
* History of or ongoing auto-immune disease
* Suffering from hemostatic disorder

Linked to infection:

* Presence of bacterial, fungal or viral infection in or close to the area of interest or treatment for these affections
* History of streptococcal illness (such as recurrent sore throat or acute articular rheumatism)
* Recurrent genital herpes (several times a year)

Linked to neoplasia:

* History of cancer in areas close to the injection site (external urogenital, anal or vaginal)
* Actual cancer or presence of pre-cancerous cells (e.g. vaginal dysplasia)

Linked to previous or ongoing treatments:

* Under treatment with aspirin, anticoagulant, platelets aggregation inhibiting drugs, NSAIDs and Vitamin C or treated within 1 week prior to inclusion
* Under local hyaluronic acid-like hydrating treatment within 4 weeks prior to inclusion
* History of hyaluronic acid injection of >14 ml in any part of the body within the last year
* History of correction with DESIRIAL® range or other resorbable implants with similar indication within 1 year prior to inclusion
* History of correction with permanent implants including fat graft or semi-permanent in the area of injection
* Surgical history on Labia Minora within one year prior inclusion
* Surgical history on Labia Majora

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients having an improvement on the Global Aesthetic Improvement Scale (GAIS) | 12 weeks
  Proportion of patients having an improvement on the GAIS, evaluated by the patient (after mirror self-examination), 12 weeks after baseline injection. 5 possible grades: 1) Very much improved, 2) much improved, 3) improved, 4) no change, 5) worse

SECONDARY OUTCOMES:
Patient self-assessed aesthetic evolution | 4 weeks, 24 weeks, 36 weeks, 52 weeks
  Patient self-assessed aesthetic evolution (after mirror self-examination) using GAIS evaluated 4, 24, 36 and 52 weeks after baseline injection. 5 possible grades: 1) Very much improved, 2) much improved, 3) improved, 4) no change, 5) worse
Patient aesthetic evolution | 4 weeks, 12 weeks, 24 weeks, 36 weeks, 52 weeks
  Patient aesthetic evolution evaluated by the Investigator (after visual observation) using GAIS evaluated 4, 12, 24, 36 and 52 weeks after baseline injection. 5 possible grades: 1) Very much improved, 2) much improved, 3) improved, 4) no change, 5) worse
Sexual function assessment | 4 weeks, 12 weeks, 24 weeks, 36 weeks, 52 weeks
  Sexual function assessment by Female Sexual Function Index (FSFI) score self-evaluated 4, 12, 24, 36 and 52 weeks after baseline injection. Auto-questionnaire with 19 multiple choice questions to measure the sexual functioning in women
Patient's satisfaction: questionnaire (PSQ) | 4 weeks, 12 weeks, 24 weeks, 36 weeks, 52 weeks
  Patient's satisfaction using a questionnaire (PSQ) evaluated 4, 12, 24, 36 and 52 weeks after baseline injection. Questionnaire with 5 questions answerable by 4 choices: not at all, a little, a lot, totally
Assessment of patient's symptoms | 4 weeks, 12 weeks, 24 weeks, 36 weeks, 52 weeks
  Assessment of patient's symptoms related to atrophy or hypotrophy of the vulvar Labia Majora (irritation/burning during daily life, irritation/burning during sport, and itching) using a Numerical Rating Scale (NRS) evaluated 4, 12, 24, 36 and 52 weeks after baseline injection. Graded scale from 0 (absent) to 10 (intolerable) in increments of 1
Patient's assessment of pain related to the injection | Baseline (injection)
  Patient's assessment of pain related to the injection, measured on a NRS during injection. Graded scale from 0 (no pain) to 10 (worst possible pain) in increments of 1
Report of adverses effects | Up to 52 weeks
  Evaluation of product safety by adverse event collection throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Fabien BOUCHER, MD, Principal Investigator
Locations (8):
- France (8):
  - Chu Henri Mondor, Créteil
  - Private office, Les Lilas
  - CHU Croix-Rousse, Lyon
  - Private office, Marseille
  - Centre de la femme, Nantes
  - Private office, Paris
  - Private office, Perpignan
  - Clinique de l'Europe, Rouen

IPD SHARING:
Plan to Share IPD: No